CLINICAL TRIAL: NCT00667056
Title: A Randomized, Double-Blind, Vehicle-Controlled, Multicenter Trial to Assess the Safety and Efficacy of 0.1% Tacrolimus Ointment in the Treatment of Chronic Allergic Contact Dermatitis
Brief Title: Study of the Safety and Efficacy of Tacrolimus Ointment in Treating Chronic Allergic Contact Dermatitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20-04-001
Record Dates: First submitted 2008-04-23; First posted 2008-04-25 (Estimated); Last update posted 2014-09-18 (Estimated); Status verified 2014-09

CONDITIONS: Dermatitis
Keywords: Chronic Allergic Contact Dermatitis; Protopic
MeSH Terms: conditions — Dermatitis | interventions — Tacrolimus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: tacrolimus ointment
- 2 (Placebo Comparator)
  Interventions: Drug: placebo ointment

INTERVENTIONS:
Drug: tacrolimus ointment — topical
  Other Names: Protopic; FK506 ointment
  Arms: 1
Drug: placebo ointment — topical
  Arms: 2

SUMMARY:
A study of subjects with a known nickel allergy comparing Tacrolimus to placebo, both associated with nickel patches to determine the safety and efficacy of treating Chronic Allergic Contact Dermatitis with Tacrolimus Ointment

ELIGIBILITY:
Inclusion Criteria:

* Subject has a history of allergy to nickel

Exclusion Criteria:

* Subject is pregnant or lactating
* Subject fails to react to the nickel disks (grade 0), reacts with a questionable (grade 1) or extreme (grade 4) reaction or the subject's reactions on the left and right arms are not of the same grade of intensity
* Subject has a known hypersensitivity to any component of the test medications
* Subject has any other significant dermatological condition that affects >10% of the body surface area or general medical condition that could interfere with the study evaluation
* Subject has any significant medical condition that could compromise immune responsiveness

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2004-07; Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Success using the Physician's Global Assessment (PGA) | 8 Weeks

SECONDARY OUTCOMES:
Investigator and subject ACD Sign and Symptoms | 8 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: use central contact, Study Director — Astellas Pharma US, Inc.
Locations (10):
- United States (10):
  - Washington D.C., District of Columbia
  - Kansas City, Kansas
  - Shawnee, Kansas
  - Louisville, Kentucky
  - New Orleans, Louisiana
  - Minneapolis, Minnesota
  - New York, New York
  - Portland, Oregon
  - Hershey, Pennsylvania
  - Lynchburg, Virginia

REFERENCES:
- [Background] Belsito D, Wilson DC, Warshaw E, Fowler J, Ehrlich A, Anderson B, Strober BE, Willetts J, Rutledge ES. A prospective randomized clinical trial of 0.1% tacrolimus ointment in a model of chronic allergic contact dermatitis. J Am Acad Dermatol. 2006 Jul;55(1):40-6. doi: 10.1016/j.jaad.2006.03.025. Epub 2006 May 26. PMID 16781290